CLINICAL TRIAL: NCT04811599
Title: Deep Learning Algorithm for the Diagnosis of Gastrointestinal Diseases Depending on Tongue Images
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Director of Qilu Hospital gastroenterology department, Shandong University
Other Study IDs: 2020-SDU-QILU-G056
Record Dates: First submitted 2021-03-20; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Gastrointestinal Disease
Keywords: Gastrointestinal Disease; tongue image; artificial intelligence; deep learning; gastrointestinal flora
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tougue coating,gastric mucosa and stool sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- deep learning algorithm group: Before patients going through colonoscopy or gastroscopy ,taking them tongue images and collecting basic information by mobile phone with Anymed.After examination,endoscopic report and histology analysis is collected .Categorizing the images by gastrointestinal diseases，developing and validating a deep learning algorithm for the diagnosis of digestive tract diseases depending on tongue images.Extracting tougue coating,gastric mucosa and stool DNA by high-throughput sequencing,and analyzing their composation,adundance and diversity.

SUMMARY:
The purpose of this study is to analysize the relationship between the characteristics of tongue image and the diagnosis of gastrointestinal diseases , then develop and validate a deep learning algorithm for the diagnosis of gastrointestinal diseases depending on tongue images, so as to improve the objectiveness and intelligence of tongue diagnosis. At the same time, gastrointestinal flora of common tongue images were analyzed in order to provide a microecological basis for understanding the relationship between tongue images and digestive tract diseases.

DETAILED DESCRIPTION:
Tongue diagnosis is an important part of traditional Chinese medicine.According to traditional Chinese medicine theory,health condition can assessed by observing tougue features,including color, gloss, shape and coating of the tongue, tongue features reflect gastric mucosal state, disease classification and prognosis. Recently, deep learning based on central neural networks (CNN) has shownTongue diagnosis is an important part of traditional Chinese medicine.According to traditional Chinese medicine theory,health condition can assessed by observing tougue features,including color, gloss, shape and coating of the tongue, tongue features reflect gastric mucosal state, disease classification and prognosis. Recently, deep learning based on central neural networks (CNN) has shown multiple potential in detecting and diagnosing gastrointestinal diseases. However, there is still a blank in recognition of gastrointestinal diseases .This study aims to develop and validate a deep learning algorithm for the diagnosis of digestive tract diseases depending on tongue images,and analyze gastrointestinal flora of common tongue images.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 - 80 years undergoing endoscopic examination;patients gave informed consent and signed informed consent.

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 - 80 years undergoing endoscopic examination
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-03-21 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
The diagnostic accuracy of gastrointestinal diseases with deep learning algorithm | 1 month
  The diagnostic accuracy of gastrointestinal diseases with deep learning algorithm.

SECONDARY OUTCOMES:
The diagnostic sensitivity of gastrointestinal diseases with deep learning algorithm | 1 month
  The diagnostic sensitivity of gastrointestinal diseases with deep learning algorithm.
The diagnostic specificity of gastrointestinal diseases with deep learning algorithm | 1 month
  The diagnostic specificity of gastrointestinal diseases with deep learning algorithm
The diagnostic positive predictive value of gastrointestinal diseases with deep learning algorithm | 1 month
  The diagnostic specificity of gastrointestinal diseases with deep learning algorithm
The diagnostic negative predictive value of gastrointestinal diseases with deep learning algorithm | 1 month
  The diagnostic specificity of gastrointestinal diseases with deep learning algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Study Chair — Study Principal investigator
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China